CLINICAL TRIAL: NCT00739843
Title: Cognitive and Functional Status and Dialysis Outcomes in Older Hemodialysis Patients
Status: Terminated | Type: Observational
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Other Study IDs: 15813B
Record Dates: First submitted 2008-08-20; First posted 2008-08-22 (Estimated); Last update posted 2016-11-01 (Estimated); Status verified 2016-10

CONDITIONS: Dementia; Cognition; End-stage Renal Disease
Keywords: Dementia,; Cognitive Disorders,; Hemodialysis
MeSH Terms: conditions — Dementia; Kidney Failure, Chronic; Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to estimate how quickly cognitive status and functional status in older patients on hemodialysis declines.

DETAILED DESCRIPTION:
Dialysis outcome measures, which predict morbidity and mortality of younger patients on renal replacement therapy, such as dialysis clearance, do not correlate with survival of the elderly patients on hemodialysis. Survival of older patients on hemodialysis is significantly worse when compared to that of the younger patients. Conditions commonly affecting older adults, such as functional decline, cognitive impairment, depression and declining quality of life have not been well studied in hemodialysis population. There may be an important relationship between these measurements and outcomes in older dialysis patients. Institution of appropriate age-specific interventions could result in improved health status and mortality of older patients on hemodialysis. Our broad objective is to better understand global functioning of the elderly dialysis patients and its possible impact on dialysis outcomes in attempt to improve health care of the older patients receiving hemodialysis.

ELIGIBILITY:
Inclusion Criteria:

* Prevalent and incident hemodialysis patients over the age of 60, receiving hemodialysis treatments at the University of Chicago outpatient dialysis program.

Exclusion Criteria:

* Patients 59 and younger, and patients with the following medical conditions: malignancies currently requiring chemotherapy or radiation therapy, severe heart failure (NYHA class IV), known HIV infection, or currently active hepatic encephalopathy.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All prevalent and incident hemodialysis patients over the age of 60, receiving hemodialysis treatments at the University of Chicago outpatient dialysis program at the time of the study will be invited to participate.
Sampling Method: Non-Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2007-11; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nicole Stankus, MD, MSc, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago Chronic Hemodialysis Centers, Chicago, Illinois, United States